CLINICAL TRIAL: NCT01665378
Title: Impact of Pre-Pregnancy Micronutrient Supplementation on Maternal and Child Outcomes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: Micronutrient Initiative (Other); The Mathile Institute for the Advancement of Human Nutrition (Other)
Responsible Party: Principal Investigator, Usha Ramakrishnan, Professor, Emory University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: IRB00051384; 10-1196-UEMORY-01 (Other: Other)
Record Dates: First submitted 2012-08-13; First posted 2012-08-15 (Estimated); Last update posted 2021-07-08 (Actual); Status verified 2021-07

CONDITIONS: Anemia; Intrauterine Growth Retardation; Preterm Delivery; Iron Deficiency
Keywords: prepregnancy; micronutrient; supplementation; maternal; child; health
MeSH Terms: conditions — Anemia; Fetal Growth Retardation; Premature Birth; Iron Deficiencies | interventions — Iron; Folic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (6):
- Multiple micronutrient - 1 (Experimental): The study population has been divided into 6 arms receiving 3 different pre-pregnancy interventions. The study uses a double blind design therefore the supplements are differentiated by a letter and a color: P/Purple, Q/Black, S/Brown, M/Green, T/Orange, H/Red. Multiple micronutrient groups 1 and 2 receive:
  Vitamin A (μg) 800 Vitamin D (IU) 600 Vitamin E (mg) 10 Vitamin C (mg) 70 Thiamine (mg) 1.4 Riboflavin (mg) 1.4 Niacin (mg) 18 Vitamin B6 (mg) 1.9 Vitamin B12 (μg) 2.6 Folic acid (μg)* 2800 Iron (mg)* 60 Zinc (mg) 15 Copper (mg) 2 Selenium (μg) 65 Iodine (μg) 150
  Interventions: Dietary Supplement: Multiple Micronutrient
- Iron and folic acid - 1 (Active Comparator): The study population has been divided into 6 arms receiving 3 different pre-pregnancy interventions. The study uses a double blind design therefore the supplements are differentiated by a letter and a color: P/Purple, Q/Black, S/Brown, M/Green, T/Orange, H/Red. Iron and folic acid groups 1 and 2 receive: iron (60mg) and folic acid (2800μg), based on current WHO recommendations for WRA.
  Interventions: Dietary Supplement: Iron and Folic Acid
- Folic Acid - 1 (Placebo Comparator): The study population has been divided into 6 arms receiving 3 different pre-pregnancy interventions. The study uses a double blind design therefore the supplements are differentiated by a letter and a color: P/Purple, Q/Black, S/Brown, M/Green, T/Orange, H/Red. Folic acid groups 1 and 2 receive: 2800 μg FA once a week during the pre-pregnancy period.
  Interventions: Dietary Supplement: Folic Acid
- Multiple Micronutrient - 2 (Experimental): The study population has been divided into 6 arms receiving 3 different pre-pregnancy interventions. The study uses a double blind design therefore the supplements are differentiated by a letter and a color: P/Purple, Q/Black, S/Brown, M/Green, T/Orange, H/Red. Multiple micronutrient groups 1 and 2 receive:
  Vitamin A (μg) 800 Vitamin D (IU) 600 Vitamin E (mg) 10 Vitamin C (mg) 70 Thiamine (mg) 1.4 Riboflavin (mg) 1.4 Niacin (mg) 18 Vitamin B6 (mg) 1.9 Vitamin B12 (μg) 2.6 Folic acid (μg)* 2800 Iron (mg)* 60 Zinc (mg) 15 Copper (mg) 2 Selenium (μg) 65 Iodine (μg) 150
  Interventions: Dietary Supplement: Multiple Micronutrient
- Iron and Folic Acid - 2 (Active Comparator): The study population has been divided into 6 arms receiving 3 different pre-pregnancy interventions. The study uses a double blind design therefore the supplements are differentiated by a letter and a color: P/Purple, Q/Black, S/Brown, M/Green, T/Orange, H/Red. Iron and folic acid groups 1 and 2 receive: iron (60mg) and folic acid (2800μg), based on current WHO recommendations for WRA.
  Interventions: Dietary Supplement: Iron and Folic Acid
- Folic acid - 2 (Placebo Comparator): The study population has been divided into 6 arms receiving 3 different pre-pregnancy interventions. The study uses a double blind design therefore the supplements are differentiated by a letter and a color: P/Purple, Q/Black, S/Brown, M/Green, T/Orange, H/Red. Folic acid groups 1 and 2 receive: 2800 μg FA once a week during the pre-pregnancy period.
  Interventions: Dietary Supplement: Folic Acid

INTERVENTIONS:
Dietary Supplement: Multiple Micronutrient — There is no current recommendation for weekly MM supplements for WRA. Therefore, we propose a supplement that contains: The same amounts of iron and folic acid as the weekly, pre-natal IFA supplement; An amount of vitamin D based on the Food and Nutrition Board's Recommended Daily Allowances (RDA); UNICEF/WHO/UNU recommended amounts of remaining nutrients (UNIMMAP recommendations). The supplement is taken weekly during pre-pregnancy.
  Vitamin A (μg) 800 Vitamin D (IU) 600 Vitamin E (mg) 10 Vitamin C (mg) 70 Thiamine (mg) 1.4 Riboflavin (mg) 1.4 Niacin (mg) 18 Vitamin B6 (mg) 1.9 Vitamin B12 (μg) 2.6 Folic acid (μg)* 2800 Iron (mg)* 60 Zinc (mg) 15 Copper (mg) 2 Selenium (μg) 65 Iodine (μg) 150
  Arms: Multiple Micronutrient - 2; Multiple micronutrient - 1
Dietary Supplement: Iron and Folic Acid — The doses of weekly and daily iron (60mg) and folic acid (2800μg) are based on current WHO recommendations for WRA.
  Arms: Iron and Folic Acid - 2; Iron and folic acid - 1
Dietary Supplement: Folic Acid — It is unethical to have a placebo group as FA is universally recommended for WRA to prevent neural tube defects. Therefore, the control group will receive 2800 μg FA once a week during the pre-pregnancy period. This dosage is safe and meets the minimum recommended intake of 400 μg/d for Women of Reproductive Age (WRA). Recent studies have shown that a weekly dose of 2800 μg FA is as effective as a daily dose of 400 μg in improving folic acid and reducing homocysteine levels among WRA.
  Arms: Folic Acid - 1; Folic acid - 2

SUMMARY:
The study evaluates the efficacy of providing weekly iron-folate (IFA) supplements or Multiple Micronutrient (MM) supplements before pregnancy in increasing birth weight and duration of gestation as well as maternal and infant iron status.

DETAILED DESCRIPTION:
Low birth weight and anemia remain intractable problems in many developing countries despite considerable efforts to address them. Intervening with just prenatal iron-folate (IFA) supplements may not be the best approach given the substantial demands for iron by maternal and fetal tissues. Therefore, there is an urgent need to evaluate the additional contribution of prepregnancy interventions.

The study evaluates the efficacy of providing weekly iron-folate (IFA) supplements or Multiple Micronutrient (MM) supplements before pregnancy in increasing birth weight and duration of gestation as well as maternal and infant iron status.

ELIGIBILITY:
Inclusion Criteria:

* 18-35 years old
* Currently married
* Currently living in one of the 10 communes and intends to live in the areas for 24 months following recruitment
* Plans to have children in the next year
* Agrees to participate with informed consent

Exclusion Criteria:

* Currently pregnant
* Delivered in the previous six months
* Regularly consumed IFA or MM supplements in the past 2 months
* Severe anemia (Hb < 7 g/L)
* History of high risk pregnancy including abruptio placenta, placenta previa, gestational diabetes, pregnancy induced hypertension, coagulation disorders, thrombocytopenia or chronic vascular, renal or systemic disease and drug use
* Chronic hematological diseases, hereditary defects of red cells or hemoglobin

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 5011 (Actual)
Dates: Start 2011-10 (Actual); Primary Completion 2014-09 (Actual); Study Completion 2019-12 (Actual)

PRIMARY OUTCOMES:
Birth Size | At birth
  Infants' weight, length and head circumference will be measured as early as possible within 24 hours after birth using standard procedures. All measurements will be obtained in duplicate by the same data collector. Weight-for-age and length-for-age z scores will be calculated using the 2006 WHO reference data.
Gestational Age | At birth
  Gestational age will be calculated based on the date of last menstrual period. This method has been shown to be reliable in previous work and we expect precise estimates since we will be visiting women weekly from baseline during the prepregnancy period and will exclude women who may be have delivered in the past 6 months.
Child growth | From birth through 24 months
  Length and weight will be measured at birth, 1, 3, 6, 9, 12, 15, 18, and 24 mo
Child development | Up to 7 years post enrollment
  Child development will be measured using the Bayley Scales for Infant Development III at 12 and 24 mo and the Wechsler Intelligence Scale for Children at age 6-7 y
Weight-for-age Z score (WAZ) | Up to 7 years post enrollment
  Weight-for-age Z score (WAZ) in offspring of women receiving only FA, offspring of women who receive weekly pre-pregnancy IFA, and offspring of women who receive weekly MM supplements
Height-for-age Z score (HAZ) | Up to 7 years post enrollment
  Height-for-age Z score (HAZ) in offspring of women receiving only FA, offspring of women who receive weekly pre-pregnancy IFA, and offspring of women who receive weekly MM supplements
Weight -for-Height Z (WHZ) or Body Mass Index Z score (BMIZ) | Up to 7 years post enrollment
  Weight -for-Height Z score (WHZ) or BMIZ in offspring of women receiving only FA, offspring of women who receive weekly pre-pregnancy IFA, and offspring of women who receive weekly MM supplements
Body composition (Lean mass/fat free mass index) | Up to 7 years post enrollment
  Body composition (Lean mass/fat free mass index) in offspring of women receiving only FA, offspring of women who receive weekly pre-pregnancy IFA, and offspring of women who receive weekly MM supplements

SECONDARY OUTCOMES:
Mothers' iron status | At baseline and 1 and 3 months post partum
  Venous blood samples (5 ml) will be collected from women at: baseline, the first prenatal visit and at 1 and 3 months post partum. Anemia will be defined as Hb value <12 g/L for non-pregnant women,and <11g/L for pregnant women and infants, and iron deficiency as serum ferritin <12 μg/L (93).
Infants' iron status | 1 and 3 months of age
  Infant iron status will be measured in cord blood samples (5 ml) obtained at delivery and at 3 months of age using a capillary blood sample (100 l) that will be obtained from a heel prick.
  The hemoglobin concentration will be measured from a drop of blood using the HEMOCUE B- Hb photometer. The blood samples will then be centrifuged and serum samples will be aliquotted into microcuvettes and handled in the same way as described for mothers. Serum ferritin and transferrin receptor concentrations will be assayed using the ELISA method.
Maternal depression | At baseline, during pregnancy, 3 months postpartum
  Center for Epidemiological Studies Depression Scale (CES-D) and Edinburgh Postnatal Depression Scale (EPDS)

CONTACTS AND LOCATIONS:
Overall Officials: Usha Ramakrishnan, PhD, Principal Investigator — Emory University
Locations (1):
- Thainguyen University of Medicine and Pharmacy, Hành Phố Thái Nguyên, Thái Nguyên, Vietnam

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Nguyen PH, Lowe AE, Martorell R, Nguyen H, Pham H, Nguyen S, Harding KB, Neufeld LM, Reinhart GA, Ramakrishnan U. Rationale, design, methodology and sample characteristics for the Vietnam pre-conceptual micronutrient supplementation trial (PRECONCEPT): a randomized controlled study. BMC Public Health. 2012 Oct 24;12:898. doi: 10.1186/1471-2458-12-898. PMID 23092451
- [Background] Nguyen PH, Gonzalez-Casanova I, Young MF, Truong TV, Hoang H, Nguyen H, Nguyen S, DiGirolamo AM, Martorell R, Ramakrishnan U. Preconception Micronutrient Supplementation with Iron and Folic Acid Compared with Folic Acid Alone Affects Linear Growth and Fine Motor Development at 2 Years of Age: A Randomized Controlled Trial in Vietnam. J Nutr. 2017 Aug;147(8):1593-1601. doi: 10.3945/jn.117.250597. Epub 2017 Jun 14. PMID 28615372
- [Result] Nguyen PH, DiGirolamo AM, Gonzalez-Casanova I, Pham H, Hao W, Nguyen H, Truong TV, Nguyen S, Harding KB, Reinhart GA, Martorell R, Ramakrishnan U. Impact of preconceptional micronutrient supplementation on maternal mental health during pregnancy and postpartum: results from a randomized controlled trial in Vietnam. BMC Womens Health. 2017 Jun 17;17(1):44. doi: 10.1186/s12905-017-0401-3. PMID 28623904
- [Result] Nguyen PH, Young M, Gonzalez-Casanova I, Pham HQ, Nguyen H, Truong TV, Nguyen SV, Harding KB, Reinhart GA, Martorell R, Ramakrishnan U. Impact of Preconception Micronutrient Supplementation on Anemia and Iron Status during Pregnancy and Postpartum: A Randomized Controlled Trial in Rural Vietnam. PLoS One. 2016 Dec 5;11(12):e0167416. doi: 10.1371/journal.pone.0167416. eCollection 2016. PMID 27918586
- [Result] Ramakrishnan U, Nguyen PH, Gonzalez-Casanova I, Pham H, Hao W, Nguyen H, Truong TV, Nguyen S, Harding KB, Reinhart GA, Neufeld LM, Martorell R. Neither Preconceptional Weekly Multiple Micronutrient nor Iron-Folic Acid Supplements Affect Birth Size and Gestational Age Compared with a Folic Acid Supplement Alone in Rural Vietnamese Women: A Randomized Controlled Trial. J Nutr. 2016 Jul;146(7):1445S-52S. doi: 10.3945/jn.115.223420. Epub 2016 Jun 8. PMID 27281806
- [Derived] Nguyen PT, Nguyen PH, Tran LM, Khuong LQ, Van Nguyen S, Young MF, DiGirolamo A, Ramakrishnan U. The Relationship of Preterm and Small for Gestational Age with Child Cognition During School-Age Years. J Nutr. 2024 Aug;154(8):2590-2598. doi: 10.1016/j.tjnut.2024.06.012. Epub 2024 Jun 25. PMID 38936548
- [Derived] Ramakrishnan U, Wimalasena ST, Young MF, Khuong LQ, Tran LM, Hoffman DJ, Martorell R, Nguyen PH. Preconception Micronutrient Supplementation Affects Maternal BMI and Body Composition Postpartum: A Randomized Controlled Trial in Vietnam. J Nutr. 2024 Apr;154(4):1440-1448. doi: 10.1016/j.tjnut.2024.02.024. Epub 2024 Feb 26. PMID 38417549
- [Derived] Duong C, Young MF, Nguyen PH, Tran L, Patel S, Ramakrishnan U. Temporal Dietary Diversity Patterns Are Associated with Linear Growth but Not Ponderal Growth in Young Children in Rural Vietnam. J Nutr. 2023 Oct;153(10):3083-3091. doi: 10.1016/j.tjnut.2023.06.030. Epub 2023 Jun 25. PMID 37364684
- [Derived] Young MF, Nguyen P, Tran LM, Khuong LQ, Martorell R, Ramakrishnan U. Long-Term Association Between Maternal Preconception Hemoglobin Concentration, Anemia, and Child Health and Development in Vietnam. J Nutr. 2023 May;153(5):1597-1606. doi: 10.1016/j.tjnut.2023.03.015. Epub 2023 Mar 15. PMID 36925072
- [Derived] Tran LM, Nguyen PH, Young MF, Ramakrishnan U, Alderman H. Home environment and nutritional status mitigate the wealth gap in child development: a longitudinal study in Vietnam. BMC Public Health. 2023 Feb 8;23(1):286. doi: 10.1186/s12889-023-15156-2. PMID 36755279
- [Derived] Nguyen PH, Young MF, Khuong LQ, Tran LM, Duong TH, Nguyen HC, Martorell R, Ramakrishnan U. Maternal Preconception Body Size and Early Childhood Growth during Prenatal and Postnatal Periods Are Positively Associated with Child-Attained Body Size at Age 6-7 Years: Results from a Follow-up of the PRECONCEPT Trial. J Nutr. 2021 May 11;151(5):1302-1310. doi: 10.1093/jn/nxab004. PMID 33693757
- [Derived] Gonzalez-Casanova I, Nguyen PH, Young MF, Harding KB, Reinhart G, Nguyen H, Nechitillo M, Truong TV, Pham H, Nguyen S, Neufeld LM, Martorell R, Ramakrishnan U. Predictors of adherence to micronutrient supplementation before and during pregnancy in Vietnam. BMC Public Health. 2017 May 16;17(1):452. doi: 10.1186/s12889-017-4379-4. PMID 28511688
- [Derived] Young MF, Hong Nguyen P, Addo OY, Pham H, Nguyen S, Martorell R, Ramakrishnan U. Timing of Gestational Weight Gain on Fetal Growth and Infant Size at Birth in Vietnam. PLoS One. 2017 Jan 23;12(1):e0170192. doi: 10.1371/journal.pone.0170192. eCollection 2017. PMID 28114316
- [Derived] Deputy NP, Nguyen PH, Pham H, Nguyen S, Neufeld L, Martorell R, Ramakrishnan U. Validity of gestational age estimates by last menstrual period and neonatal examination compared to ultrasound in Vietnam. BMC Pregnancy Childbirth. 2017 Jan 11;17(1):25. doi: 10.1186/s12884-016-1192-5. PMID 28077098
- [Derived] Young MF, Nguyen PH, Addo OY, Hao W, Nguyen H, Pham H, Martorell R, Ramakrishnan U. The relative influence of maternal nutritional status before and during pregnancy on birth outcomes in Vietnam. Eur J Obstet Gynecol Reprod Biol. 2015 Nov;194:223-7. doi: 10.1016/j.ejogrb.2015.09.018. Epub 2015 Sep 28. PMID 26454228